CLINICAL TRIAL: NCT02610309
Title: Family-based Crisis Intervention With Suicidal Adolescents in the Emergency Department: A Randomized Clinical Trial
Brief Title: Family-based Crisis Intervention With Suicidal Adolescents in the ED
Acronym: FBCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Elizabeth Wharff, Clinical Researcher, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P00000105
Record Dates: First submitted 2015-11-13; First posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Suicide
Keywords: family-based crisis intervention; adolescent suicide
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family-Based Crisis Intervention (Experimental): The Family-Based Crisis Intervention (FBCI) is a single-session intervention that takes place in the Emergency Department. Adolescents randomized to the experimental condition received a standard psychiatric evaluation followed by the experimental intervention. FBCI was administered by licensed psychiatric social workers who were trained in the intervention. The research clinician provided FBCI to the suicidal adolescent and his/her parent(s)/guardian(s) in a 60-90 minute session in which she helped the adolescent and family develop a joint crisis narrative of the problem and taught them cognitive-behavioral skill-building, therapeutic readiness, psycho-education about depression, and safety planning.
  Interventions: Behavioral: Family-Based Crisis Intervention
- Treatment As Usual (No Intervention): Treatment as usual included an emergency psychiatry evaluation (standard care).

INTERVENTIONS:
Behavioral: Family-Based Crisis Intervention — This intensive ED-based intervention with suicidal adolescents and their families includes cognitive behavioral skill building, psychoeducation, enhancing therapeutic readiness, safety planning, and co-creation of a joint crisis narrative.
  Arms: Family-Based Crisis Intervention

SUMMARY:
The Family Based Crisis Intervention (FBCI) is an emergency psychiatry intervention designed to sufficiently stabilize suicidal adolescents within a single ED visit so that they may return home safely with their families. This study is a randomized clinical trial of FBCI v. TAU in an urban Emergency Department.

DETAILED DESCRIPTION:
In current practice, treatment as usual (TAU) for suicidal adolescents includes evaluation, with little or no intervention provided in the Emergency Department (ED), and disposition, usually to an inpatient psychiatry unit. The Family Based Crisis Intervention (FBCI) is an emergency psychiatry intervention designed to sufficiently stabilize suicidal adolescents within a single ED visit so that they may return home safely with their families. The intervention works intensively with both the adolescent and the family, so that the caregiver has the knowledge and skills to help the adolescent after discharge.

In this study, suicidal adolescents (ages 13-18) and their families presenting for psychiatric evaluation to a large pediatric ED were randomized to receive FBCI or treatment as usual (TAU). Patients and caregivers completed self-report measures of suicidality, family empowerment, and satisfaction with care provided at pre-test, post-test, and 3 follow up time-points over a one-month period. Clinicians contacted the adolescent and caregiver at these timepoints to administer the questionnaires and assure safety planning was being carried out.

ELIGIBILITY:
Inclusion Criteria:

* adolescent presenting to the ED with suicidality
* presence of a consenting parent or legal guardian with whom the adolescent resided.

Exclusion Criteria:

* either adolescent or parent/guardian lacked fluency in English;
* adolescent was not medically stable, including intoxication;
* adolescent demonstrated cognitive limitations prohibiting completion of research instruments;
* adolescent presented with active psychosis;
* adolescent required physical or medication restraint in the ED.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 143 (Actual)
Dates: Start 2012-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Disposition at discharge from the ED (psychiatric hospitalization or other) | one day, one week, and one month
  The primary outcome measure is disposition (psychiatric hospitalization vs. less restrictive level of care) after receiving the FBCI intervention or TAU. Psychiatric hospitalization was reassessed at 1 day, 1 week and 1 month intervals after randomization.

SECONDARY OUTCOMES:
Family Empowerment Scale (FES) | one month
  The FES is a 34-item self-report instrument designed to measure the level of empowerment in parents/guardians of a child/adolescent with emotional difficulties. Based upon a bi-dimensional definition of perceived and expressed empowerment, the FES contains three separate subscales: family, community/political, and service system. The FES demonstrates good reliability (internal consistency alpha values of .88, .87, and .88 on each of the three subscales). Validity of the FES subscales has been supported by multi-rater classification of items by expert panelists (inter-rater kappa coefficients of agreement yielded values of .83, .77, and .73 for each of the three subscales) as well as strong evidence of known-groups validity.15 The parents/guardians completed the FES at post-test, 3 day, 1 week, and one month timepoints.
Client Satisfaction Questionnaire (CSQ-8) | one day
  The CSQ-8 is an 8 item questionnaire that was developed to assess global client satisfaction. Items assess quality of service received, kind of service received, willingness to recommend to a friend, amount of help received, overall satisfaction, and willingness to come back for future service. Participants responded using a 4-point Likert scale scored from 1 to 4, and total scores range from 8 to 32. Higher scores indicate greater satisfaction. The parent/guardian completed the CSQ-8 as part of the post-test only.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Wharff, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States